CLINICAL TRIAL: NCT02160496
Title: A Randomized Study to Assess the Effect of Diets With Different Protein Composition - Mainly Coming From Lean Red Meat - in Body Weight and Lipid Profile in Overweight and Obese Women
Brief Title: A Study to Assess the Effect of Diets With Different Protein Composition - Mainly Coming From Lean Red Meat - in Body Weight and Lipid Profile in Overweight and Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Aragones de Ciencias de la Salud (Other Government)
Responsible Party: Principal Investigator, Fernando Civeira, Professor, Instituto Aragones de Ciencias de la Salud
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEICA;PI13/00108; I+CS-HUMS-B80_PI13/00108 (Other: I+CS-HUMS-B80)
Record Dates: First submitted 2014-06-05; First posted 2014-06-10 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Weight Loss; Obesity; Overweight; Diet, Reducing; Lipids
Keywords: Weight Loss; Obesity; Overweight; Diet, Reducing; Lipids
MeSH Terms: conditions — Weight Loss; Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- 20% protein hypocaloric diet (Active Comparator): Participants were advised with a hypocaloric diet with the following composition: 20% protein, 30% fat and 50% carbohydrates. A wide variety of healthy foods typically coming from a mediterranean diet and specific exercise recommendations are provided to the subjects.
  Interventions: Behavioral: Weight loss interventional study with 20% protein-diet
- 27% protein hypocaloric diet (Active Comparator): Participants were advised with a hypocaloric diet with the following composition: 27% protein, 30% fat and 43% carbohydrates. A wide variety of healthy foods typically coming from a mediterranean diet and specific exercise recommendations are provided to the subjects.
  Interventions: Behavioral: Weight loss interventional study with 27% protein-diet
- 35% protein hypocaloric diet (Active Comparator): Participants were advised with a hypocaloric diet with the following composition: 35% protein, 30% fat and 35% carbohydrates. A wide variety of healthy foods typically coming from a mediterranean diet and specific exercise recommendations are provided to the subjects.
  Interventions: Behavioral: Weight loss interventional study with 35% protein-diet

INTERVENTIONS:
Behavioral: Weight loss interventional study with 20% protein-diet
  Arms: 20% protein hypocaloric diet
Behavioral: Weight loss interventional study with 27% protein-diet
  Arms: 27% protein hypocaloric diet
Behavioral: Weight loss interventional study with 35% protein-diet
  Arms: 35% protein hypocaloric diet

SUMMARY:
The objective of the study is to assess the effect of diets with different protein composition (20%, 27% and 35%), mainly coming from animal proteins such as lean red meat, on body weight and lipid profile in overweight and obese women. A dietary intervention is carried out during 3 months in 90 women who are individually randomized to an hypocaloric diet with three types of macronutrient composition: 1) 35% proteins, 30% fat and 35% carbohydrates; 2) 27% proteins, 30% fat and 43% carbohydrates and 3) 20% proteins, 30% fat and 50% carbohydrates. Around 50% of total proteins in diet come from lean red meat (leg or shoulder of lamb) by providing up to 15 different recipes to participants to use them as part of the diet. At the beginning of the study, after 6 weeks and at the end of the intervention, the following parameters are determined: anthropometric (weight, waist circumference, body mass index and body composition), blood pressure, dietary (72-hours dietary registry) and exercise assessments and biochemical analysis (total cholesterol, triglycerides, HDL cholesterol, LDL cholesterol, apolipoprotein A1, apolipoprotein B, iron, transferrin, ferritin, uric acid, glucose, HbA1c, insulin and adipokines). In 3-months visit, participants will be advised to follow the prescribed diets during the next 3 months. Monitoring visits with the nutritionist will not be performed. A follow-up visit will be done after 3-months of end of intervention (at 6-months after beginning the study) to assess the long-time efficacy on main endpoint of each diet. In this visit only anthropometric parameters (weight, waist circumference, body mass index and body composition) will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years old.
* Body mass index between 27.5 - 40.
* Steady weight in last 3 months (±3 kg).
* Informed consent provided.

Exclusion Criteria:

* Presence of uncontrolled endocrinological pathology (including hypothyroidism).
* Type 2 diabetes mellitus with bad metabolic control (HbA1c > 8%).
* Lipid-lowering drugs in the last 3 months.
* Intake of functional foods with plant sterols in the past 6 weeks.
* Vitamin supplements intake.
* Hormone replacement therapy.
* Consumption of Orlistat in the last 2 months
* High intake of alcohol (> 30 gr./day).
* Any serious disease which involves less than 1 year life expectancy or, in investigators judgment, limit the follow-up of an homogeneous diet throughout the study.
* Pregnancy or intention of pregnancy during the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in body weight and lipid profile of diets with different protein composition in overweight and obese women.. | After 3 months of intervention
  The main outcome is to study the effect of diets with different protein composition (20%, 27% and 35%), mainly coming from lean red meat, on body weight and lipid profile in overweight and obese women.

SECONDARY OUTCOMES:
Change in body composition (by including waist circumference, fat mass and muscle mass) of diets with different protein composition in overweight and obese women. | After 3 months of intervention.
Change in carbohydrates metabolism of diets with different protein composition in overweight and obese women. | After 3 months of intervention.

OTHER OUTCOMES:
Change in blood pressure of diets with different protein composition in overweight and obese women. | After 3 months of intervention.
Change in body weight of diets with different protein composition in overweight and obese women.. | After 3 months of study completion (at 6-months after beginning the study)
  In 3-months visit, participants will be advised to follow the prescribed diets during the next 3 months. Monitoring visits with the nutritionist will not be performed. A follow-up visit will be done after 3-months of end of intervention (at 6-months after beginning the study) to assess the long-time efficacy on main endpoint of each diet. In this visit only anthropometric parameters (weight, waist circumference, body mass index and body composition) will be determined.
Change in adipokines concentration of diets with different protein composition in overweight and obese women. | After 3 months of study completion.
  In 3-months visits serum plasma, adipokines concentration will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Civeira, MD, PhD, Principal Investigator — Unidad de Lípidos/Laboratorio de Investigación Molecular; Hospital Universitario Miguel Servet; Instituto Aragonés de Ciencias de la Salud (Zaragoza, Spain); Rocio Mateo-Gallego, MSc, Principal Investigator — Unidad de Lípidos/Laboratorio de Investigación Molecular; Hospital Universitario Miguel Servet; Instituto Aragonés de Ciencias de la Salud (Zaragoza, Spain)

REFERENCES:
- [Derived] Mateo-Gallego R, Lamiquiz-Moneo I, Perez-Calahorra S, Marco-Benedi V, Bea AM, Baila-Rueda L, Laclaustra M, Penalvo JL, Civeira F, Cenarro A. Different protein composition of low-calorie diet differently impacts adipokine profile irrespective of weight loss in overweight and obese women. Nutr Metab Cardiovasc Dis. 2018 Feb;28(2):133-142. doi: 10.1016/j.numecd.2017.10.024. Epub 2017 Nov 4. PMID 29329923
- [Derived] Mateo-Gallego R, Marco-Benedi V, Perez-Calahorra S, Bea AM, Baila-Rueda L, Lamiquiz-Moneo I, de Castro-Oros I, Cenarro A, Civeira F. Energy-restricted, high-protein diets more effectively impact cardiometabolic profile in overweight and obese women than lower-protein diets. Clin Nutr. 2017 Apr;36(2):371-379. doi: 10.1016/j.clnu.2016.01.018. Epub 2016 Jan 29. PMID 26875447